CLINICAL TRIAL: NCT03820778
Title: Whole Body MRI to Identify Atypical Neurofibromas in Patients With NF1 and High Plexiform Neurofibroma Tumor Burden
Brief Title: Whole Body MRI to Identify Atypical Neurofibromas in Patients With NF1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Miriam Bornhorst, Assistant Professor Division of Oncology and Center for Genetics Medicine, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00010431
Record Dates: First submitted 2019-01-04; First posted 2019-01-29 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Neurofibromatosis 1; Neurofibroma; Atypical Neurofibroma; Atypical Neurofibromatosis; Plexiform Neurofibroma; Von Recklinghausen Disease
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma; Neurofibromatosis, type 4, of Riccardi; Neurofibroma, Plexiform

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study Arm (Experimental): Whole Body MRI along with standard of care regional MRI and blood draw at enrollment followed by Whole Body MRI along with standard of care regional MRI and blood draw after 4-6 months.
  Interventions: Diagnostic Test: Whole Body MRI

INTERVENTIONS:
Diagnostic Test: Whole Body MRI — WBMRI with axial and coronal STIR (short inversion time inversion recovery) images + DWI (diffuse weighted imaging) will be performed and compared to regional MRI to assess value of this diagnostic test for the identification of suspicious looking lesions (i.e. diffuse nodular lesions or atypical plexiform neurofibroma)

SUMMARY:
This study is being conducted to determine if Whole Body MRI (WBMRI) can be used to identify Atypical Neurofibromas (ANF) in Neurofibromatosis Type 1 (NF1) patients with high tumor burden. Each enrolled participant will have two (2) WBMRIs without sedation during the study period. Eligible participants must be Male or Female between the ages of 8-30 with diagnosed NF1; with one or more PN greater than 3cm in diameter and willing to comply with study procedures.

DETAILED DESCRIPTION:
This is a study to determine the feasibility of using Whole Body MRI (WBMRI) to detect Atypical Plexiform Neurofibromas (ANF) among Neurofibromatosis Type 1 (NF1) patients who are at highest risk for developing these tumors. In order to do this, the investigators will prospectively obtain WBMRI scans on patients with high plexiform tumor burden (which investigators will define as >=1 plexiform neurofibroma (PN) that is >3cm in diameter on MRI) at the same time as their regularly scheduled MRI to allow for radiographic comparison of the identified PNs. In this study, the investigators will plan to establish a method that effectively characterizes PNs in terms of their volume, radiographic appearance on WBMRI and association with clinical characteristics.

As an exploratory aim, the investigators plan to collect blood samples from each patient at the same time as the MRI to determine the feasibility of isolating cfDNA (circulating free DNA) from plasma of patients with high plexiform tumor burden.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 8-30 years of age
2. Confirmed diagnosis of NF1
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Prior MRI documentation confirming >=1 PN that is >3cm in diameter

Exclusion Criteria:

1. Unable to undergo MRI without sedation
2. Presence of metal or other devices that are contraindicated for MRI

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
To determine if WBMRI can be used to identify ANF in NF1 patients with high tumor burden. | 2-3 years
  Number of NF1 participants with high tumor burden who have ANF on WBMRI

SECONDARY OUTCOMES:
Determine if clinical signs and symptoms correlate with tumor burden and/or the presence of ANF on WBMRI | 2-3 years
  Number of patients with high PN tumor burden who have clinical symptoms

OTHER OUTCOMES:
Determine if the cfDNA levels correlate with presence of ANF. | 3-4 years
  Level of cfDNA in plasma of participants with ANF compared to participants without ANF

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Bornhorst, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen R, Dombi E, Widemann BC, Solomon J, Fuensterer C, Kluwe L, Friedman JM, Mautner VF. Growth dynamics of plexiform neurofibromas: a retrospective cohort study of 201 patients with neurofibromatosis 1. Orphanet J Rare Dis. 2012 Oct 4;7:75. doi: 10.1186/1750-1172-7-75. PMID 23035791
- [Background] Kim A, Stewart DR, Reilly KM, Viskochil D, Miettinen MM, Widemann BC. Malignant Peripheral Nerve Sheath Tumors State of the Science: Leveraging Clinical and Biological Insights into Effective Therapies. Sarcoma. 2017;2017:7429697. doi: 10.1155/2017/7429697. Epub 2017 May 16. PMID 28592921
- [Background] Higham CS, Dombi E, Rogiers A, Bhaumik S, Pans S, Connor SEJ, Miettinen M, Sciot R, Tirabosco R, Brems H, Baldwin A, Legius E, Widemann BC, Ferner RE. The characteristics of 76 atypical neurofibromas as precursors to neurofibromatosis 1 associated malignant peripheral nerve sheath tumors. Neuro Oncol. 2018 May 18;20(6):818-825. doi: 10.1093/neuonc/noy013. PMID 29409029
- [Background] Beert E, Brems H, Daniels B, De Wever I, Van Calenbergh F, Schoenaers J, Debiec-Rychter M, Gevaert O, De Raedt T, Van Den Bruel A, de Ravel T, Cichowski K, Kluwe L, Mautner V, Sciot R, Legius E. Atypical neurofibromas in neurofibromatosis type 1 are premalignant tumors. Genes Chromosomes Cancer. 2011 Dec;50(12):1021-32. doi: 10.1002/gcc.20921. Epub 2011 Aug 24. PMID 21987445
- [Background] Mautner VF, Asuagbor FA, Dombi E, Funsterer C, Kluwe L, Wenzel R, Widemann BC, Friedman JM. Assessment of benign tumor burden by whole-body MRI in patients with neurofibromatosis 1. Neuro Oncol. 2008 Aug;10(4):593-8. doi: 10.1215/15228517-2008-011. Epub 2008 Jun 17. PMID 18559970
- [Background] Dominguez-Vigil IG, Moreno-Martinez AK, Wang JY, Roehrl MHA, Barrera-Saldana HA. The dawn of the liquid biopsy in the fight against cancer. Oncotarget. 2017 Dec 8;9(2):2912-2922. doi: 10.18632/oncotarget.23131. eCollection 2018 Jan 5. PMID 29416824
- [Background] Plotkin SR, Bredella MA, Cai W, Kassarjian A, Harris GJ, Esparza S, Merker VL, Munn LL, Muzikansky A, Askenazi M, Nguyen R, Wenzel R, Mautner VF. Quantitative assessment of whole-body tumor burden in adult patients with neurofibromatosis. PLoS One. 2012;7(4):e35711. doi: 10.1371/journal.pone.0035711. Epub 2012 Apr 27. PMID 22558206
- [Background] Ahlawat S, Fayad LM, Khan MS, Bredella MA, Harris GJ, Evans DG, Farschtschi S, Jacobs MA, Chhabra A, Salamon JM, Wenzel R, Mautner VF, Dombi E, Cai W, Plotkin SR, Blakeley JO; Whole Body MRI Committee for the REiNS International Collaboration; REiNS International Collaboration Members 2016. Current whole-body MRI applications in the neurofibromatoses: NF1, NF2, and schwannomatosis. Neurology. 2016 Aug 16;87(7 Suppl 1):S31-9. doi: 10.1212/WNL.0000000000002929. PMID 27527647
- [Background] Cai W, Kassarjian A, Bredella MA, Harris GJ, Yoshida H, Mautner VF, Wenzel R, Plotkin SR. Tumor burden in patients with neurofibromatosis types 1 and 2 and schwannomatosis: determination on whole-body MR images. Radiology. 2009 Mar;250(3):665-73. doi: 10.1148/radiol.2503080700. PMID 19244040
- [Background] Wasa J, Nishida Y, Tsukushi S, Shido Y, Sugiura H, Nakashima H, Ishiguro N. MRI features in the differentiation of malignant peripheral nerve sheath tumors and neurofibromas. AJR Am J Roentgenol. 2010 Jun;194(6):1568-74. doi: 10.2214/AJR.09.2724. PMID 20489098